CLINICAL TRIAL: NCT04880369
Title: DAGMAR: Phytoestrogens and Breast Cancer - Effects of Phytoestrogens on Markers of Disease Progression and Gene Expression
Brief Title: Phytoestrogens and Breast Cancer - Effects of Phytoestrogens on Markers of Disease Progression and Gene Expression
Acronym: DAGMAR
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Disapproved by relevant Danish ethical committee
Sponsor: Danish Cancer Society (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Cecilie Kyrø, Principal Investigator, Danish Cancer Society
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R174-A11507-17-S52
Record Dates: First submitted 2021-05-05; First posted 2021-05-10 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer; Breast Neoplasms; Breast Cancer Female
Keywords: Phytoestrogens; Isoflavones; Lignans; Gene expression; Breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Soybean Proteins; Lignans

STUDY DESIGN:
Intervention Model Description: The study planned to include 150 women.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Lignan capsule (Experimental): 1 capsule/day from baseline to end-of-follow-up (approx. 4 months)
  Interventions: Dietary Supplement: Lignans
- Isoflavones capsule (Experimental): 1 capsule/day from baseline to end-of-follow-up (approx. 4 months)
  Interventions: Dietary Supplement: Soy isoflavones
- Placebo capsule (Placebo Comparator): 1 capsule/day from baseline to end-of-follow-up (approx. 4 months)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Soy isoflavones — Commercially available dietary supplement (capsule) containing 60 mg isoflavones (genistein, daidzein and glycitein).
  Arms: Isoflavones capsule
Dietary Supplement: Lignans — Commercially available dietary supplement (capsule) containing 63 mg lignans (secoisolaricirecinol)
  Arms: Lignan capsule
Dietary Supplement: Placebo — The placebo capsules are supplied and packaged by Region Hovedstadens Apotek (Denmark) and will contain lactose monohydrate, potato starch, gelatin, magnesium stearate and talc.
  Arms: Placebo capsule

SUMMARY:
The aim is to investigate if soy isoflavones and lignans affect markers of disease progression and gene expression among breast cancer patients receiving neo-adjuvant treatment in a three arm, double-blinded, randomized placebo-controlled trial (RCT) comparing: soy isoflavone supplementation, lignan supplementation, and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with breast cancer at "Brystkirurgisk Afdeling" at Rigshospitalet and Herlev Hospitals (within the last 30 days).
* Advised (and accepted) to receive neo-adjuvant treatment
* Primary unilateral breast cancer
* Treatment is expected to be curative
* Is expected to be able to attend surgery

Exclusion Criteria:

* Allergic to soy
* Celiac disease
* Inflammatory bowel disease
* Not understanding Danish (patient material and questionnaires are in Danish)
* Prior diagnosis of breast cancer
* Use of dietary supplements containing lignans or isoflavones three months prior to diagnosis

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Ki-67 | Change from baseline (diagnosis of breast cancer) to end-of-study (surgery): Approx. four months (neo-adjuvant setting)
  Ki-67 can be measured using immunohistochemistry (IHC) and using the transcript from gene expression data (see secondary outcomes). As the latter is superior and less biased, the Ki-67 based on the transcript will be used as primary measure of Ki67.

SECONDARY OUTCOMES:
Apoptosis marker caspase-3 | Change from baseline (diagnosis of breast cancer) to end-of-study (surgery): Approx. four months (neo-adjuvant setting)
Proliferation Index | Change from baseline (diagnosis of breast cancer) to end-of-study (surgery): Approx. four months (neo-adjuvant setting)
  Based on expression data from 79 genes encoding proliferative and cell cycle markers. Gene expression will be analyzed using a microarray (GeneChip® Human Genome U133 Plus 2.0 Array, Affymetrix, USA)
Patient reported outcomes | Change for completion of first questionnaire (shortly after diagnosis) to second questionnaire (close to time of surgery). Approx. four months (neo-adjuvant setting)
  Well-being

OTHER OUTCOMES:
Fecal microbiome: | Change measured in first fecal sample (shortly after diagnosis) to second fecal sample (close to time of surgery). Approx. four months (neo-adjuvant setting)
  The microbial community composition will be characterized using the 16sRNA method (Illumina MiSeq Platform).

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon approval from relevant authorities and in accordance with the law
Supporting Information: Study Protocol, SAP, ICF
Access Criteria: Please request this information from PI Cecilie Kyrø, Ceciliek@cancer.dk